CLINICAL TRIAL: NCT03845673
Title: Randomized Trial Comparing Two Fiber Regimens for the Reduction of Symptoms of Constipation
Brief Title: Fiber Regimens for Constipation Symptoms
Acronym: constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Clifford Wai, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0703-457
Record Dates: First submitted 2011-08-02; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Constipation
Keywords: Bowel recipe; Bristol stool form scale; Konsyl; psyllium; wheat bran
MeSH Terms: conditions — Constipation | interventions — Psyllium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psyllium (Experimental): This group of patients was given psyllium for 6 weeks
  Interventions: Dietary Supplement: Psyllium
- Bowel recipe (Experimental): This group was administered a specialized bowel recipe for 6 weeks
  Interventions: Dietary Supplement: Bowel recipe

INTERVENTIONS:
Dietary Supplement: Psyllium — Psyllium fiber (Konsyl; Konsyl Pharmaceuticals, Easton, Md)
  Arms: Psyllium
Dietary Supplement: Bowel recipe — consisted of 1 cup of unprocessed wheat bran, 1 cup of applesauce, and 1/4 cup of prune juice.
  Arms: Bowel recipe

SUMMARY:
The objective of the current study is to compare the effects of bowel recipe with psyllium on symptoms associated with constipation.

DETAILED DESCRIPTION:
Patients presenting to the urogynecology clinics at Parkland Health and Hospital System and UT Southwestern Medical Center at Dallas from July 2003 to July 2005 were screened for symptoms of constipation. Subjects were randomized to a 6-week course of either psyllium (Konsyl, Konsyl Pharmaceuticals, Easton, MD) or a special bowel recipe. The bowel recipe was a modification of that used by Behm and consisted of 1 cup of unprocessed wheat bran, 1 cup of applesauce, and 1/4 cup of prune juice. A validated constipation scoring questionnaire12 was administered to participants at the beginning and at the end of the six-week study period. During the six-week trial patients also kept a bowel diary recording characteristics of each bowel movement.

ELIGIBILITY:
Inclusion Criteria:

* fluent and literate in either English or Spanish.
* responds affirmatively to at least two symptoms according to Rome II criteria for functional constipation, for at least 12 weeks

Exclusion Criteria:

* pregnant or less than six weeks postpartum
* six weeks post abdominal surgery,
* colostomy
* history of bowel obstruction, inflammatory bowel disease, diagnosis of slow colonic transit time, spinal cord injury, neurogenic disease, myopathic disorders, or cognitive impairment, history of an allergic reaction to psyllium or any of the ingredients contained in the bowel recipe, such as wheat bran, prunes, or apples.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2003-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Constipation questionnaire scores | 6 weeks
  A validated constipation scoring questionnaire was administered to participants at the beginning and at the end of the 6-week study period. Previous studies have shown that dietary modifications can result in significant improvement in constipa- tion scores and symptom relief as early as 2 to 6 weeks. The questionnaire consisted of 8 variables: (i) frequency of bowel movements, (ii) painful evacuation, (iii) incomplete evacuation, (iv) abdominal pain, (v) length of time per attempt, (vi) assis- tance with defecation, (vii) unsuccessful attempts at evacuation per 24 hours, and (viii) duration of constipation. Each variable was scored on a range of 0 to 4 (except for ''assistance for defecation,'' which was scored from 0 to 2), and a cumulative score was determined. A global score of 0 is generally considered normal, and a maximum score of 30 indicates severe con- stipation.

SECONDARY OUTCOMES:
frequency of bowel movements | 6 weeks
  number of bowel movements per week

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Y Wai, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States